CLINICAL TRIAL: NCT03854877
Title: DagisWork - Improved Health Behaviour and Wellbeing: a Randomized Controlled Workplace Intervention
Brief Title: DagisWork-a Workplace Health Behaviour E-intervention
Acronym: DagisWork
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: University of Helsinki (Other); University of Jyvaskyla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FinnishIOH
Record Dates: First submitted 2017-09-14; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-08

CONDITIONS: Health Behavior
Keywords: Health behaviour; Work place intervention; Stress; Physical activity; Nutrition; e-health; Mindfulness
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster randomized two group behavioral intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health behaviour intervention (Experimental): Personalised health behaviour e-health intervention. The intervention uses the principles of acceptance-commitment therapy (ACT). It aims to promote health habits. Based on personal needs participants can choose tasks for physical activity, relaxation, healthy eating, sleep etc. They get regular feedback, tasks and support from their personal trainer via phone and computer.
  Interventions: Behavioral: Health behaviour intervention
- Control group (No Intervention): Only before and after measurements

INTERVENTIONS:
Behavioral: Health behaviour intervention — The intervention uses the principles of acceptance-commitment therapy (ACT). It aims to increase healthy eating and good sleep. Based on personal needs participants can choose task for physical activity, relaxation, healthy eating, sleep eg. Their get regular feedback and support from their personal trainer via phone and computer.
  Arms: Health behaviour intervention

SUMMARY:
The main aim of the study is to test effectiveness of a multiple intervention program aimed at making positive changes to health behaviour and stress. Effectiveness of a 4 month workplace intervention, with virtual coaching and co-worker-support, will be assessed as changes in subjective and objective measures of stress, work ability, recovery and health behaviour.

DETAILED DESCRIPTION:
Consequences of psychosocial stress can be seen in personnel's health such as long lasting imbalance between consumptive and restoring physiological processes (allostatic load, AL) that increase the risk of physical diseases and mental health problems and poor health behaviours. Chronic work stress induces adverse emotional and physical responses, which are triggered by perception of demands that exceed the person's capacity to cope (Folkman et al. 1986).

Health behaviour can be improved both by increasing personnel's' resources and removing stress-causing factors (Lamontagne et al. 2007). Mindfulness based cognitive therapy aims at increasing stress resources by developing emotional and behavioral experiences. It combines aspects of cognitive approach including dialectic behavior therapy and Acceptance and Commitment Therapy (ACT). Mindfulness and acceptance-based interventions have positive consequences for physical activity and quality of life (Kangasniemi et al. 2015, Khoury et al. 2015). Novel results suggest that the approach is effective to reduce work stress also (Aikens et al. 2014). A four month intervention with virtual life habit coaching, individualised exercises and mindfulness-based techniques will be performed. The aim is to achieve significant and long lasting changes in life habits and stress of employees.

The extensive measurements including both self-evaluated and objective measurements together with multifaceted viewpoint provide profound knowledge of occupational health. They also create a comprehensive picture of preschool setting as an arena for healthy lifestyle and well-being. A new issue is the concert of different kinds of work load factors, and their interacting role in biomarkers for work stress. If proven effective, the health behaviour intervention tested in preschool environment, can be modified to suit also other occupational settings. The health economic evaluation, together with aforementioned measurement, offer information for different stakeholders on whether interventions are economically worthwhile for participating municipalities and occupational health care. The results of study are beneficial also for policy-makers in different sectors.

Aims and hypotheses Primary hypotheses

1. The intervention has a positive effects on long-term physiological adaptation to stress, biological health risk factors, recovery, and sickness absences among personnel.
2. The interventions directly enhance personnel's health behavior including eating habits, physical activity and experienced stress.

Secondary hypotheses

1. The physiological change in stress regulating systems caused by work related factors (psychosocial, cognitive, and physical) is associated with personnel's change health risk load (AL) and recovery.
2. Subjective psychological and cognitive factors of stress, recovery and even mental health symptoms are individually related to physiological responses, which can be characterized more precisely by the combined assessment of hormonal, neuronal responses and new methods of system biology.
3. The intervention will have positive economic effect (costs and benefits).
4. The intervention will have positive changes in self-efficasy

ELIGIBILITY:
Inclusion Criteria:

* Voluntary
* Working in municipal city of Espoo or Kouvola in preschool

Exclusion Criteria:

* Pregnancy
* Retirement during the intervention

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Allostatic load (AL) | Change from baseline in stress after four months
  Allostatic load (AL) (allostatic load and allostatic overload refers to the cumulative result of an allostatic state) is measured by the following primary and secondary markers: salivary cortisol (µg/dl) heart rate variability measurement [RMSSD, (ms)], (hsCRP (mg/l), HbA1c (mmol/mol), triglycerides (mmol/l). Salivary cortisol is the mean of morning and evening samples (Aardal, E.&Holm, A. 1995), (RMSSD is the value on recovery during sleeping (First_beat Manual 2014). Clinical cutoff values are used for salivary cortisol, hsCRP, HbA1c and triglycerides and age-reference value (HUSLAB Manual 2018). All markers are dichotomized (0 = below the clinical or age-reference; 1= exceeds the clinical or age-reference). Total Allostatic load is calculated as the sum of all measures (range 0 to 5) (Altman et. al.1986). Total Allostatic load we shown before and after the intervention.
Perceived stress | Change from baseline in stress after four months
  General Health Questionnaire (GHQ-12). The scale includes 12 items. The four response choices (0 "Not at all", 1 "Same as usual", 2 "Rather more than usual" and 3 "Much more than usual") will be dichotomized as follows: 1=0, 2=1, 3=2, 4=3. GHQ-12 case ≥ 3 points (range 0-36). The higher values indicate higher psychological symptoms. The reference mean value is 10.3 (SD 5.0) points (Holi, Marttunen, Aalberg 2003).

SECONDARY OUTCOMES:
Economic benefits | Sickness absence absence [ (Time Frame: approx. 3 years (from 2016 to 2019) ]
  Length (1-365 days/year) of sickness absence and frequency of sickness absence episodes (i.e. frequency of all sickness absence periods within year) obtained from employer records, including dates of absence due to sickness without medical cause information.
Intuitive eating | Change from baseline after four months
  The Intuitive Eating Scale, 21-items. All items are rated on a five point Likert-scale (1 totally disagree, 5 totally agree). The sum of all items indicates the level of eating habits. Higher values indicate better eating habits.
Eating habits | Change from baseline after four months.
  The three factor eating questionnaire-R 18 (TFEQ-18). All items of the three factors (cognitive restraint, uncontrolled eating, emotional eating) are rated on a four point Likert- scale (1 definitely true, 4 definitely false). Higher values indicate higher cognitive restraint, uncontrolled eating and emotional eating.
Measured physical activity | Change from baseline after four months
  Accelerometer. Average number of steps per week, at least five days and 10 hours data/day. The program counts the physical activity time in different levels (inactive, light, moderate and heavy). The higher number of steps indicate higher physical activity as well as the moderate or heavy activity.
Work ability | Change from baseline after four months
  Question on the current Work Ability (WA) compared with the lifetime best is assessed using one item with a response scale from 0 not able to work at all to 10, my best work ability ever. The result are reported as mean and classification. The higher value is better work ability (Seitsamo et al. 2011).
Cognitive failures at work | Change from baseline after four months
  Workplace cognitive failure scale (WCFS) (Wallace & Chen, 2005). The 15 items of the scale are rated on a 5-point scale (1 =never to 5=several times per day) and sum up to total WCF. All items are summed -up to total WCFS. The higher value indicates more cognitive failures.
Self-efficacy | Change from baseline after four months
  The Self-efficacy beliefs questionnaire (Scharzer & Renner 2000). External and internal attribute. The scale are rated on a 5-point scale (1 =never to 5=several times per day). All items are summed-up.
Sleep | Change from baseline after four months
  The Jenkins sleep questionnaire. Four items of the scale are rated on a 6-point scale (1= never to 6 = every night). All items are summed-up. The higher value means more problems in sleeping (Jenkins et al 1988).

CONTACTS AND LOCATIONS:
Overall Officials: Sampsa Puttonen, PhD, Principal Investigator — Finnish Institute of Occupational Health
Locations (1):
- Finnish Institute of Occupational Health, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karihtala T, Puttonen S, Valtonen AM, Kautiainen H, Hopsu L, Heinonen A. Role of physical activity in the relationship between recovery from work and insomnia among early childhood education and care professionals: a cross-sectional study. BMJ Open. 2024 Mar 19;14(3):e079746. doi: 10.1136/bmjopen-2023-079746. PMID 38508638